CLINICAL TRIAL: NCT04427696
Title: The Effect of Walking Exercise on Sleep Quality in Sedentary Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Feifei Wang (Other)
Responsible Party: Sponsor-Investigator, Feifei Wang, Principal Investigator, Eotvos Lorand University
Organization: Eotvos Lorand University (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 2018/421
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Walking; Sleep; Stress, Psychological; Lifestyle, Sedentary; Life Change Events
MeSH Terms: conditions — Stress, Psychological; Sedentary Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic walking (Active Comparator): The participants in this arm were obligated to carry out one hour aerobic walking (goal setting walking) daily. The goal of aerobic walking: 1. at least 60 steps per minute; 2. continuously walking for 10 minutes.
  Interventions: Behavioral: Aerobic walking intervention
- No aerobic walking (Placebo Comparator): The participants in this arm were requested to maintain sedentary life, without joining other physical exercise programmes.
  Interventions: Behavioral: Aerobic walking intervention

INTERVENTIONS:
Behavioral: Aerobic walking intervention — Walking exercise is self-controlled and tracked by daily dairy. All of the participants are obligated to record the start and end time of walking every day. And pedometers will be used for tracking walking steps including heart rate and calories. We plan to use pedometer in our study, which was reported the most accurate pedometer and suitable for scientific research. For the ones who are in the control group, they have to keep sedentary lifestyle, and no regular walking exercise, and they are agree to be in the comparable members in our study.

SUMMARY:
The primary goal of this study is to examine the effect of one-hour walking exercise on sleep quality in adults. The second goal of this study is to explore a feasible exercise method to promote sleep quality to all age groups, in order to improve sleep quality in overall population. The study attempts to unfold how the daily exercise, such as walking, benefits sleep quality. This study hypothesis that one-hour walking improves sleep quality in general population.

DETAILED DESCRIPTION:
In order to test the hypothesis that walking exercise improves sleep quality in general population, the investigators conducted a randomized (case-control) cross-over trial. The targeted population is the physically and mentally healthy adults (18+). The health status was self-reported, the investigators did not organize physical and mental examination for participants in this study. The investigators recruited participants both online and off-line. The call-for-participants advertisement distributed in social media platforms such as Facebook, WeChat etc.

There were two groups in this study: walking group, and control group. The call-for-participants advertisement was distributed through online platforms and by posters. In the advertisement, all people were welcomed to participate, after receiving the applications, the investigators assessed the participant. In order to test the hypothesis that walking exercise improve sleep quality in general population, the investigators conducted a randomized (case-control) cross-over trial.

Participants can only be accepted after approval from the research team who performed the group discussion and evaluation of the sedentary behavior. If the participants meet the sedentary criteria, the participants would be informed the consent and terms and conditions to participate the study. Participants were randimzed into two groups by lottery (intervention and control group). The first phase intervention lasted for four weeks. At the beginning and at end of the intervention, the investigators assessed the sleep quality of participants by the Pittsburgh Sleep Quality Index (PSQI), Perceived Stress Scale (PSS) and Satisfaction With Life Scale (SWLS). The second phase was a wash period (4-week) and the third phase was a 4-week intervention. It has to be noted that at the beginning of the third phase, the participants in the two groups exchanged their role to receive active interventions. Participants in each group were coded by an autonomous number with characters.

Walking exercise was self-controlled and tracked by daily dairy and pedometers. All of the participants are obligated to record the start and end time of walking every day. And pedometers (mode: Omron HJ-112) were used for tracking walking steps including heart rate, calories and miles. For the ones who were in the control group, they had to keep sedentary lifestyle.

The participants had the responsibility to carry out the walking practice every day in the first and third phase. Every participant was counselled and gave their written informed consent before entering into the trial. The participation of this project was voluntary, unpaid. During the trial, all participants were free to quit the project with reasonable reasons, the investigators will not force anyone to continue the project if they cannot insist on. The investigators would inform the results of the first phase if the participant requests.

ELIGIBILITY:
Inclusion Criteria:

* between 18-60 years old
* without physical or metal diseases

Exclusion Criteria:

* People who responded to join the study were screened either online or face-to-face by two principal questions: 1: Do you participate in any kind of regular exercise programs (weight-lifting, walking, running, swimming etc.)? 2. Are you involved in any physical or sport teams? If the respondent answered "Yes" to at least one of the questions, he/she would be excluded from the study because it could interfere with the effect of intervention.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-05-26 (Actual)

PRIMARY OUTCOMES:
Sleep quality | 12 weeks
  Sleep quality is measured by Pittsburgh Sleep Quality Index, the score of which ranges from 0 to 21. If the score is less than 5, it indicates good sleeper, otherwise, it will be indicated as poor sleeper. Overall, higher score, poorer sleep quality.
Stress | 12 weeks
  Stress is measured by Perceived Stress Scale . Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
Life satisfaction | 12 weeks
  Life satisfaction is assessed by Satisfaction With Life Scale. Participants indicate how much they agree or disagree with each of the 5 items using a 7-point scale that ranges from 7 strongly agree to 1 strongly disagree.

SECONDARY OUTCOMES:
Height | 12 weeks
  cm
Weight | 12 weeks
  kg

CONTACTS AND LOCATIONS:
Locations (1):
- Feifei Wang, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No
There is not plan for making IPD available to other researchers, as it has been confirmed in the consent form. What we can share is the result of the whole intervention study and intervention process.